CLINICAL TRIAL: NCT04073186
Title: Evaluation of A Marketed Silicone Hydrogel Spherical Lens Used for Monovision Correction of Presbyopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-6349
Record Dates: First submitted 2019-08-28; First posted 2019-08-29 (Actual); Results first posted 2021-05-18 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Visual Acuity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ACUVUE® OASYS with Transitions™ (Experimental): Eligible subjects between the ages of 40 to 70 years of age and habitual wearers of soft contact lenses will be fitted with the study lens for two wearing cycles.
  Interventions: Device: ACUVUE® OASYS with Transitions™

INTERVENTIONS:
Device: ACUVUE® OASYS with Transitions™ — JJVC Marketed Contact Lens

SUMMARY:
This is a single-masked, dispensing clinical trial. A total of approximately 48 myopic and 32 hyperopic eligible subjects will be targeted to complete the study. Subjects will be fit in the study lens, optimized if required and worn for approximately 2 weeks. Subjects will then have a washout period of approximately 1 week and be refit in the lenses and be dispensed for an additional 2 weeks of wear.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all the following criteria to be enrolled in the study:

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. The subject must be between 40 and 70 years of age at the time of screening.
  4. Subjects must own a wearable pair of spectacles if required for their distance vision.
  5. The subject must be an adapted monovision soft contact lens wearer in both eyes (i.e., worn lenses a minimum of 2 days per week for at least 8 hours per wear day, for 1 month of more duration).
  6. The subject's distance spherical equivalent refraction must be in the range of +3.50 D to -4.00 D in each eye.
  7. The subject's refractive cylinder must be ≤1.00 D in each eye.
  8. The subject's ADD power must be in the range of +0.75 D to +2.50 D.
  9. The subject must have best corrected distance visual acuity of 20/20-3 or better in each eye.

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently Pregnant or lactating.
  2. Any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, recurrent herpes simplex/zoster, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g., hepatitis, tuberculosis).
  3. Use of any of the following medications within 1 week prior to enrollment: oral retinoid isotretinoin (e.g. Accutane), oral tetracyclines, oral phenothiazines (e.g., Haldol, Mellaril, Thorazine, Elavil, Pamelor, Compazine), systemic steroids.
  4. Any previous, or planned, ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, lid procedures, cataract surgery, retinal surgery, dacryocystorhinostomy, etc.).
  5. Use of any ocular medication, with the exception of rewetting drops.
  6. Participation in any contact lens or lens care product clinical trial within 7 days prior to study enrollment.
  7. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
  8. Any known hypersensitivity or allergic reaction to OPTI-FREE® Puremoist® care cleaning solution, non-preserved rewetting drop solution or sodium fluorescein.
  9. History of herpetic keratitis.
  10. Entropion, ectropion, chalazia, glaucoma, history of recurrent corneal erosions.
  11. A history of amblyopia, strabismus or binocular vision abnormality.
  12. Clinically significant (Grade 3 or 4) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
  13. Any ocular infection or inflammation.
  14. Any ocular abnormality that may interfere with contact lens wear.
  15. Any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - VRC-East, Jacksonville, Florida
  - Advanced Eyecare, Raytown, Missouri
  - Manhattan Vision Associates, New York, New York
  - Western Reserve Vision Care, Inc., Beachwood, Ohio
  - Dr. David W. Ferris & Associates, Warwick, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 91 subjects were enrolled in this study. Of those enrolled, 86 subjects were dispensed a least one study lens while 5 subjects failed to meet all eligibility criteria. Of those dispensed, 79 subjects completed the study, while 7 were discontinued.
Groups:
- Test: Subjects received the Test lens throughout the study. Subjects wore the Test lens twice for a period of approximately 2 weeks each.
Period: First Wearing Cycle
Arm/Group | Test
Started | 86
Completed | 80
Not Completed | 6
Not completed — Time required to complete last two study visits exceeds study deadline | 1
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1
Not completed — Lens Discomfort | 2
Not completed — Unsatisfactory Visual Response due to Test Article | 1
Period: Second Wearing Cycle
Arm/Group | Test
Started | 80
Completed | 79
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Test
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.8 (6.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 13
  White | 67
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 86

OUTCOME MEASURES:

1. Primary Outcome: Vision Scores
Description: Vision Scores were assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: 2-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation impacting a primary endpoint.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Test (First Wearing Cycle): All subjects that wore the Test lens during the first wearing cycle
- Test (Second Wearing Cycle): All subjects that wore the Test lens during the second wearing cycle
Arm/Group | Test (First Wearing Cycle) | Test (Second Wearing Cycle)
Number analyzed (Participants) | 76 | 76
Units on a Scale | 59.38 (19.700) | 56.19 (23.387)
Statistical Analysis 1: Comparison: Test (First Wearing Cycle); Test type: Superiority — The superiority of the First wearing Cycle was concluded if the lower confidence limit of leastsquare mean as greater than 32; Linear Mixed Model; the Kenward and Roger method was used for the denominator degrees of freedom; Least-square Mean = 59.3, 95% CI 2-sided [54.6 to 64.0], Standard Error of Mean 2.37

2. Primary Outcome: Visual Performance (logMAR)
Description: Binocular visual performance on logMAR (Logarithm of Minimal Angle of Resolution) scale was evaluated at distance (4 meters), intermediate (64 centimeters) and near (40 centimeters) under high luminance high contrast lighting condition using ETDRS (Early Treatment Diabetic Retinopathy Study) charts. The room illuminance was required to be etween 7.3 and 7.9 EV (394-597 lux). For Distance (4 meters), the acceptable range for the chart luminance was 10.5-10.7 EV (181-208 cd/m2). For Intermediate (64 cm) and Near (40cm), the acceptable range for the chart luminance 10.8-11.1 EV (223-274 cd/m2).
  Letter-by-letter results calculated the visual performance score for each chart read. logMAR scores closer to zero, or below zero, indicate a better visual acuity. A logMAR visual performance score of 0.0 is equivalent to Snellen visual acuity of 20/20.
Time Frame: 2-Week Follow-up
Population: Subjects that completed all study visits without a major prtocol deviation impacting a primary endpoint
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Test (First Wearing Cycle) | Test (Second Wearing Cycle)
Number analyzed (Participants) | 76 | 76
logMAR
  Distance (4 Meter) | -0.08 (0.097) | -0.08 (0.100)
  Intermediate (64 CM) | -0.02 (0.096) | -0.03 (0.095)
  Near (40 CM) | 0.04 (0.085) | 0.02 (0.081)
Statistical Analysis 1: Comparison: Test (First Wearing Cycle); Test type: Superiority — The superiority of the Test lens was concluded if the upper confidence limit of least-square mean was below the pre-defined threshold 0.10 logMAR; Linear Mixed Model — Distance (4 Meter); The Kenward and Roger Method was used for the demoninator degrees of freedom; Least-square Mean = -0.084, 95% CI 2-sided [-0.124 to -0.044], Standard Error of Mean 0.0191
Statistical Analysis 2: Comparison: Test (First Wearing Cycle); Intermediate (64 CM); Test type: Superiority — The superiority of the Test lens was concluded if the upper confidence limit of least-square mean was below the pre-defined threshold 0.17 logMAR; Linear Mixed Model; The Kenward and Roger Method was used for the demoninator degrees of freedom; Least-square Mean = -0.028, 95% CI 2-sided [-0.068 to 0.012], Standard Error of Mean 0.0191
Statistical Analysis 3: Comparison: Test (First Wearing Cycle); Near (40 CM); Test type: Superiority — [test comment as in outcome 2, analysis 2]; Linear Mixed Model; The Kenward and Roger Method was used for the demoninator degrees of freedom; Least-square Means = 0.037, 95% CI 2-sided [-0.003 to 0.077], Standard Error of Mean 0.0191

3. Secondary Outcome: CLUE Vision Comparison Between First Wearing Cycle and Second Wearing Cycle
Description: Vision Scores wwere assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: Up to 2-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation impacting a primary endpoint.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Test (First Wearing Cycle) | Test (Second Wearing Cycle)
Number analyzed (Participants) | 76 | 76
Units on a Scale | 59.38 (19.700) | 56.19 (23.387)
Statistical Analysis 1: Comparison: Test (First Wearing Cycle) vs Test (Second Wearing Cycle); Test type: Superiority — The superiority of the Test lens at 4-week followup compared to it at 2-week follow-up will beconcluded if the lower confidence limit of leastsquare mean difference is greater than 0; Linear Mixed Model; the Kenward and Roger method was used for the denominator degrees of freedom; Least-square Mean Difference = -4.1, 95% CI 2-sided [-8.1 to -0.1], Standard Error of Mean 2.03 — LSM difference was calculated as Second Wearing Cycle minus First Wearing Cycle

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Approximately 1 month per subject.
Arm/Group | Test
All-Cause Mortality (participants affected / at risk) | 0/86
Serious Adverse Events (participants affected / at risk) | 1/86
Other Adverse Events (participants affected / at risk) | 0/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test (N=86)
Chest Pain (Cardiac disorders) | 1 (1) — Not related to study treatment, subject was discontinued and AE was resolved by the end of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-03): https://cdn.clinicaltrials.gov/large-docs/86/NCT04073186/Prot_SAP_000.pdf